CLINICAL TRIAL: NCT07280754
Title: Evaluation of 25(OH)D3 and LL-37 Levels in Peri-implant Sulcus Fluid in Peri-implant Diseases
Brief Title: Evaluation of 25(OH)D3 and LL-37 Levels in Periimplant Sulcus Fluid
Status: Not yet recruiting | Type: Observational
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Melek Beder, Doctor, Recep Tayyip Erdogan University
Other Study IDs: Recep Tayyip Erdogan U
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Peri Implantitis; Peri Implant Mucositis
Keywords: LL-37; peri-implanter sulcus fluid; peri-implantitis; vitamin D
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy group: Criteria such as absence of clinical signs of inflammation in the tissues, absence of bleeding on probing, PPD ≤5.0 mm, and absence of bone loss greater than 2 mm after initial healing will be sought.
- peri-implant mucositis: Criteria such as clinical signs of inflammation (erythema, swelling, suppuration) in the tissues, bleeding on probing, and an PPD of 5.0 mm will be sought. At the time of implant placement, the height of the surrounding soft tissue influences the initial probing depth.
- periimplantitis: Bleeding, inflammation, redness, edema, suppuration, and in addition to these, bone loss >5 mm and radiographically observed in PPD are observed in the tissues.

SUMMARY:
Despite technological advances that have significantly improved dental implant osseointegration and survival rates, biological complications such as peri-implantitis and peri-implant mucositis are common around the implant. The active form of vitamin D, 1,25-dihydroxyvitamin D3 (1,25(OH)2D3), can be induced by the expression of leucine-lysine-37 (LL-37), a human antimicrobial peptide in the cathelicidin family. Studies have shown that 1,25(OH)2D3 and its precursor, 25(OH)D3, significantly reduce inflammation by suppressing the release of receptor activator nuclear factor kappa b ligand (RANKL), tumor necrosis factor-alpha (TNF-α), interleukin (IL)-1, and IL-6, and by preventing alveolar bone loss. To date, many cytokines have been investigated in peri-implant sulcus fluid (PIOS). The lack of a direct study investigating vitamin D and LL-37 levels in PIOS constitutes the unique value of this project. This study aims to compare LL-37 and 25(OH)D3 levels in PIOS and examine their correlation with markers such as IL-6, IL-10, and MMP-8, as well as clinical parameters. Volunteers aged 18-65 who have received dental implants at the Recep Tayyip Erdoğan University Faculty of Dentistry and have been using their implant-supported prosthesis for at least one year and who have been informed about this study will be included in the study. The groups will be formed as peri-implant health, peri-implant mucositis, and peri-implantitis. The implants of the patients included in the study will be evaluated for probed pocket depth (PPD), clinical attachment level (CAL), suppuration (S), modified gingival index (mGI), plaque index (mPI), bleeding index (mBI), keratinized gingival amount, and attached gingival amount. PIOS and serum samples will be obtained from patients, and their relationship to periodontal status and each other will be statistically evaluated.

This project may help discover new biomarkers that can be used in the early diagnosis of peri-implantar diseases. This study could contribute to earlier treatment, lower patient costs, and even the development of new treatment plans for these diseases.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Having dental implants and using implant-supported prostheses for at least one year,
* Not having used systemic and/or topical antibiotics/anti-inflammatory drugs or mouthwashes in the last three months,
* Not having received periodontal/peri-implant treatment in the last six months.

Exclusion Criteria:

* Having a systemic disease or condition that affects peri-implant status,
* Having a metabolic bone disease,
* Bruxism,
* Being pregnant or lactating,
* Having received periodontal/peri-implant treatment within the last 6 months,
* Smoking and alcohol use,
* Taking vitamin D supplements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The G*Power analysis performed to determine the number of samples to be included in the study determined that a total of 72 samples/implants should be included, with a minimum of 24 in each group, when the power of the test was taken as 0.85, the effect size as 0.4, and the Type-1 error (α) as 0.05.
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth (PPD) | baseline
  The distance from the gingival margin to the pocket base around the implants was measured in mm using a periodontal probe, at six locations for each implant. The average value will be determined for each implant circumference.
clinical attachment level (CAL) | baseline
  Similar to the PPD measurement, this will be done by determining the distance between the pocket base and the implant neck.

SECONDARY OUTCOMES:
25-Hydroxy Vitamin D3 ((25(OH)D3)) | baseline
  25(OH)D3 levels in PIOS samples will be analyzed by ELISA or CMIA methods.
leucine leucine-37 (LL-37) | baseline
  LL-37 levels in PIOS samples will be evaluated by ELISA method.